CLINICAL TRIAL: NCT03681483
Title: A Phase 1 Trial of RO5126766 (CH5126766) in Patients With Advanced KRAS-Mutant Lung Adenocarcinomas
Brief Title: RO5126766 for Patients With Advanced KRAS-Mutant Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Chugai Pharma USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-285
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: RO5126766 (CH5126766); KRAS-Mutant; 18-285
MeSH Terms: interventions — RO5126766

STUDY DESIGN:
Intervention Model Description: Single arm, open label, multi-institution study of RO5126766 (CH5127566) in patients with KRAS mutant NSCLC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RO5126766 (CH5126766) (Experimental): The study will begin with a standard 3+3 design. The study will enroll 3 patients at the previously identified MTD15 (4mg two times per week on days 1 and 4). The period of evaluation for dose limiting toxicity will be through completion of cycle 1. If ≤1 of the 3 initial patients at the proposed dose experience a DLT, then 3 additional patients will be enrolled for a total of 6 planned patients at that dose level. Otherwise, 3 patients will be enrolled at dose level -1. If ≤ 1 of these patients experience a DLT, then 3 additional patients will be enrolled at the same dose level. If more than 1 patient experiences a DLT in dose level -1, the study will be terminated.
  Interventions: Drug: RO5126766

INTERVENTIONS:
Drug: RO5126766 — RO5126766 (CH5126766) is given 4mg twice weekly (Day 1 and Day 4 of each week) and should be taken by mouth on an empty stomach, either one hour before or two hours after a meal.
  Other Names: (CH5126766)

SUMMARY:
The purpose of this study is to test the safety of RO5126766 at different doses to find out what effects, if any, it has on people with advanced lung cancer who have previously received treatment with a PD-1 or PD-L1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of advanced NSCLC
* Documented presence of KRAS mutation
* Prior treatment with a PD-1/L1 inhibitor. Patients who were deemed not eligible for therapy with a PD-1/L1 inhibitor by their treating physician will also be eligible in the dose expansion phase.
* Prior treatment with chemotherapy
* Able to take oral medications
* Measurable and/or evaluable disease (RECIST 1.1) indicator lesion not previously irradiated
* Karnofsky performance status (KPS) ≥ 70% (ECOG of 0 or 1 also acceptable)
* Age≥ 18 years old
* Hematological and biochemical indices within the ranges shown below Hematological and biochemical indices within the ranges shown below (These measurements must be performed within two weeks [Day 14 to Day 1] before the patient is entered into the trial).

  * AST, ALT ≤ 2.5 x ULN - Total bilirubin ≤ 1.5 x ULN -Albumin≥2.5g/dL
  * Creatinine < 1.5 x ULN OR calculated creatinine clearance ≥50mL/min
  * Absolute neutrophil count (ANC) ≥ 1,200 cells/mm3
  * Hemoglobin ≥9.0 g/dL
  * Platelets ≥100,000/mm^3.
* A negative serum pregnancy test obtained within two weeks prior to the administration of the study drug in all women of child bearing potential

Exclusion Criteria:

* Patients with symptomatic brain metastasis requiring escalating doses of steroids
* Patients with grade 2 or greater diarrhea prior to study initiation despite maximal medical management
* History of any bowel disease including abdominal fistula, gastro-intestinal perforation
* History of acute pancreatitis within 1 year of study entry or history of chronic pancreatitis
* History of or ongoing alcohol abuse that, in the opinion of the treating physician, would compromise compliance or impart excess risks associated with study participation.
* Pregnant or lactating women
* Any type of systemic therapy (chemotherapy or experimental drugs) within 3 weeks of starting treatment on protocol (within 6 weeks for for nitrosoureas and mitomycin C)
* Radiotherapy within 2 weeks of starting treatment on protocol
* Prior treatment with MEK, RAF, or ERK inhibitor(s)
* Significant uncontrolled or active cardiovascular disease, specifically including, but not restricted to:

  * History of clinically significant (as determined by the treating physician) atrial arrhythmia
  * Any ventricular arrhythmia
  * History of congenital long QT syndrome.
  * Abnormal QTc (≥ 450 msec in males and ≥ 470 msec in females)
  * Ejection fraction ≤ 50% as assessed by echocardiogram
  * Concurrent congestive heart failure
  * Prior history of class III/ IV heart failure (New York Heart Association [NYHA]
  * Myocardial infarction within the last 6 months
  * Unstable angina or severe obstructive pulmonary disease
* Patients with baseline risk factors for central serous retinopathy or retinal vein occlusion such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure >21 mmHg Uncontrolled hypertension (Diastolic blood pressure > 100 mmHg; Systolic blood pressure > 150 mmHg).
* History of central serous retinopathy or retinal vein occlusion
* History of prior malignancy within 2 years that requires/ed treatment. Patients who are considered NED from a malignancy may be considered on a case by case basis.
* Known active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infections
* Patients exposed to CYP3A4 inhibitors within 7 days prior to the first dose and CYP3A4 inducers 7 days prior to the first dose. RO5126766 (CH5126766) is metabolised mainly by CYP3A4 therefore concomitant administration of strong inhibitors and inducers of cytochrome p450 3A4 enzymes is forbidden during study treatment (for a complete list please see Appendix A).
* Any other condition that, in the opinion of the investigator, may compromise the safety, compliance of the patient, or would preclude the patient from successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) | 1 year
  will be defined as the highest dose level at which ≤ 1 of 6 patients experienced a DLT.The NCI Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE) will be used to grade toxicities during the trial. DLTs are defined as any toxicity occurring during the first cycle of treatment (i.e. 4 weeks), excluding toxicites clearly related to disease progression or disease-related processes.
overall response rate (dose expansion) | 1 year
  by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Miami Cancer Institute, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm